CLINICAL TRIAL: NCT00521820
Title: A Randomized, Double-Blind, Comparator-Controlled Study of Pioglitazone HCl vs Glyburide in the Treatment of Subjects With Type 2 (Non-Insulin Dependent) Diabetes Mellitus and Mild to Moderate Congestive Heart Failure
Brief Title: Safety Comparison of Pioglitazone and Glyburide in Type 2 Diabetes Subjects With Mild to Moderate Congestive Heart Failure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Higher incidence of hospitalization for congestive heart failure in pioglitazone-treated subjects compared to glyburide treated subjects.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-00-TL-OPI-504; U1111-1114-1029 (Registry Identifier: WHO)
Record Dates: First submitted 2007-08-25; First posted 2007-08-28 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — Pioglitazone; Glyburide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone QD (Experimental)
  Interventions: Drug: Pioglitazone
- Glyburide QD (Active Comparator)
  Interventions: Drug: Glyburide

INTERVENTIONS:
Drug: Pioglitazone — Pioglitazone 30 mg (titrated to 45mg with tolerance), tablets, orally once daily and glyburide placebo-matching tablets, orally, once daily for up to 24 weeks.
  Other Names: Actos; AD-4833
  Arms: Pioglitazone QD
Drug: Glyburide — Pioglitazone placebo-matching tablets, orally, once daily and glyburide 10 mg (titrated to 15mg with tolerance), capsules, orally, once daily for up to 24 weeks.
  Arms: Glyburide QD

SUMMARY:
The purpose of this study is to compare the safety of Pioglitazone, once daily (QD), to Glyburide in Type 2 Diabetes Subjects with Mild to Moderate Congestive Heart Failure

DETAILED DESCRIPTION:
Approximately 16 million people in the United States have been diagnosed with type 2 diabetes, a prevalence rate of approximately 6%, and the numbers are expected to increase with the increasing age of the general population. The risk factors associated with development of type 2 diabetes, such as age, obesity, and diet and exercise habits, also contribute to the development of cardiovascular disease. Additionally, patients with diabetes are at an increased risk for development of microvascular and macrovascular disease.

With regard to congestive heart failure, the risk of congestive heart failure is increased in subjects with diabetes in the absence of coronary artery disease; in subjects with diabetes and established coronary artery disease there is a higher overall risk and greater risk for more severe congestive heart failure. There is evidence that increasing insulin sensitivity and reducing hyperinsulinemia may reduce cardiovascular risks by reducing blood pressure, improving endothelial function, and through cardiac remodeling and function.

Pioglitazone is a thiazolidinedione for the treatment of type 2 diabetes, and is an agonist of the peroxisome proliferator-activated receptor. Pioglitazone received marketing approval in the United States in 1999. As part of the approval process, Takeda fulfilled a postmarketing study evaluating the effects of pioglitazone in the treatment of type 2 diabetes in subjects with congestive heart failure in a6-month clinical study.

An independent Data Safety Monitoring Board used to monitor the overall safety pattern of the study and to conduct unblinded reviews of data found a difference in the composite endpoint of time to first event that approached nominal statistical significance in favor of glyburide. As a result, the committee recommended that Takeda terminate the trial. Consistent with regulatory agency requirements, Takeda is submitting an abbreviated report that focuses on the safety data derived from the terminated study.

ELIGIBILITY:
Inclusion Criteria

* Females of childbearing potential must be using appropriate birth during the entire duration of the study or must be surgically sterile.
* Subjects with a clear diagnosis of type 2 diabetes mellitus using diagnostic criteria of the American Diabetes Association who have been taking a sulfonylurea and/or insulin for at least 30 days prior to Visit 1 or who have been withdrawn from metformin therapy, during the 30 days prior to Visit 1, due to congestive heart failure.
* Subjects with a clinical diagnosis of congestive heart failure, New York Heart Association Class II or early Class III. Subjects should not previously have been in Class IV heart failure.
* Diagnosis of left ventricular congestive heart failure as evidenced by a left ventricular ejection fraction less than 40% at screening based on an echocardiogram.
* Subjects who have demonstrated the need for oral hypoglycemic agents and have participated in dietary counseling.
* Glycosylated hemoglobin greater than 7.0% at screening.
* Subjects on optimal therapy for congestive heart failure. Medication doses should be stable for at least two weeks prior to randomization.

Exclusion Criteria

* Naïve to antidiabetic therapy.
* Within the past three months were treated with rosiglitazone, pioglitazone HCl, or troglitazone or those previously treated with rosiglitazone, pioglitazone HCl, or troglitazone but discontinued from therapy due to lack of efficacy or clinical or laboratory signs of intolerance.
* Type 1 (insulin-dependent) diabetes mellitus or a history of ketoacidosis.
* Has taken any other investigational drug during the 30 days prior to Visit 1 or who will receive such a drug during the timeframe of this study.
* History of chronic alcoholism or drug abuse during the six months prior to the study.
* Has had any of the following within three months prior to Visit 1: myocardial infarction, coronary angioplasty or bypass graft, unstable angina pectoris, transient ischemic attacks, or documented cerebrovascular accident that in the investigator's opinion would warrant exclusion from the study.
* Abdominal, thoracic, or vascular surgery during the three months prior to Visit 1 that in the investigator's opinion would warrant exclusion from the study.
* Subjects with a planned surgical or catheterization intervention within the six months following Visit 1.
* Subjects awaiting cardiac transplantation.
* Intercurrent illness severe enough to require hospitalization during the three weeks prior to Visit 1.
* Body mass index greater than 48 kg/m2 as calculated by [Weight (kg)/Height (m)2].
* Anemia having a hemoglobin less than 10.5 g/dL for males and less than 10 g/dL for females.
* Thyroid stimulating hormone greater than 3.5 mU/L or less than 0.3 mU/L. The thyroid stimulating hormone can be repeated at two months. The subject is eligible if the screening thyroid stimulating hormone is elevated, and the repeat value at two months is less than 3.5 mU/L.
* Triglyceride level greater than 500 mg/dL.
* Clinical evidence of active liver disease or alanine transaminase levels greater than 1.5 times the upper limit of normal.
* Serum creatinine greater than 2.0 mg/dL for males and greater than 1.8 mg/dL for females or urinalysis protein (albumin) excretion greater than 2 plus on Combistix or equivalent (if elevated, may be re-screened in one month).
* Unstable coronary syndromes which in the opinion of the investigator would warrant exclusion from the study.
* Systolic blood pressure of greater than 150 mmHg or diastolic blood pressure greater than 100 mmHg.
* Serious uncontrolled cardiac rhythm disturbances which in the opinion of the investigator would warrant exclusion from the study.
* Symptomatic orthostatic hypotension or systolic blood pressure less than 90 mm/Hg.
* Severe, advanced peripheral vascular disease (limb threatening ischemia) or claudication resulting in the inability to walk greater than 1 block or to climb 10 stairs without interruption.
* Lower extremity amputation.
* Any other serious disease or condition at screening or at randomization which might affect life-expectancy or make it difficult to successfully manage and follow the subjects according to the protocol.
* Unexplained clinically significant findings on chest x-ray.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2000-06; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Progression of Congestive Heart Failure. | At First Event.

SECONDARY OUTCOMES:
Change from baseline in Glycosylated Hemoglobin. | Weeks 12, 20 and Final Visit.
Change from baseline in Fasting Plasma Glucose. | At All Visits.
Change from baseline in Triglycerides. | Weeks 8, 16 and Final Visit.
Change from baseline in cholesterol (total cholesterol, high-density lipoprotein and low-density lipoprotein). | Weeks 8, 16 and Final Visit.
Change from baseline in 6 Minute Walking test distance | At Final Visit
Physician & Subject Congestive Heart Failure Global Assessment Score | At Final Visit
Change in New York Heart Association classification | At All Visits.
Minnesota Living with Heart Failure Questionnaire total score. | At Final Visit.
Changes in blood pressure and heart rate. | At All Visits.
All cause mortality. | At First Event.

CONTACTS AND LOCATIONS:
Overall Officials: VP Clinical Science Strategy, Study Director — Takeda Global Research and Developmnet Center Inc

REFERENCES:
- [Result] Giles TD, Miller AB, Elkayam U, Bhattacharya M, Perez A. Pioglitazone and heart failure: results from a controlled study in patients with type 2 diabetes mellitus and systolic dysfunction. J Card Fail. 2008 Aug;14(6):445-52. doi: 10.1016/j.cardfail.2008.02.007. Epub 2008 May 27. PMID 18672190
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI